CLINICAL TRIAL: NCT00002316
Title: Phase I Study to Evaluate the Safety and Tolerance of RMP-7 Administered With Amphotericin B to Patients With HIV Infection and Cryptococcal Meningitis
Brief Title: The Safety and Effectiveness of RMP-7 Plus Amphotericin B in Patients With HIV and Cryptococcal Meningitis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alkermes, Inc. (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: Double | Purpose: Treatment
Other Study IDs: 131A; ALK01-006
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1994-12

CONDITIONS: Meningitis, Cryptococcal; HIV Infections
Keywords: AIDS-Related Opportunistic Infections; Meningitis; Drug Therapy, Combination; Antifungal Agents; Acquired Immunodeficiency Syndrome; Amphotericin B
MeSH Terms: conditions — Meningitis, Cryptococcal; HIV Infections; AIDS-Related Opportunistic Infections; Meningitis; Acquired Immunodeficiency Syndrome | interventions — RMP 7; Amphotericin B

INTERVENTIONS:
Drug: Lobradimil
Drug: Amphotericin B

SUMMARY:
To evaluate the safety of escalating doses of RMP-7 administered in persons with HIV infection and cryptococcal meningitis and to determine the MTD of the drug. To evaluate the pharmacokinetics, including cerebrospinal fluid (CSF) penetration, of amphotericin B when administered with RMP-7.

DETAILED DESCRIPTION:
Patients receive intravenous RMP-7 added to conventional therapy with intravenous amphotericin B (with or without flucytosine). Treatment continues for 14 days, with follow-up visits 4 and 12 weeks later.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Up to 1 mg/kg amphotericin B for the current episode of cryptococcal meningitis.

Patients must have:

* HIV infection.
* Acute cryptococcal meningitis.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Cardiovascular disorders including congestive heart failure, uncontrolled hypertension (seated diastolic blood pressure > 95 mm Hg), or symptomatic ischemic heart disease (angina).
* Orthostatic hypotension, defined as a decrease in systolic blood pressure of >= 20 mm Hg upon standing.
* Coma.
* Other CNS disease (e.g., other intracranial infections) that may interfere with assessment of response.
* Opening CSF pressure >= 350 mm or papilledema. (For patients with recurrent disease, evidence of mass effect on either MRI or CT excludes.)
* Any concurrent disease that would preclude participation in the study.

Patients with the following prior conditions are excluded:

* History of any bleeding disorder.
* History of active renal or hepatic disease.
* Myocardial infarction within the previous 3 months.
* Stroke within the previous 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (11):
- United States (11):
  - Los Angeles County - USC Med Ctr, Los Angeles, California
  - UCI Med Ctr, Orange, California
  - UCSD Treatment Ctr, San Diego, California
  - Univ of Kansas School of Medicine, Wichita, Kansas
  - SUNY / Health Sciences Ctr at Stony Brook, Stony Brook, New York
  - Duke Univ Med Ctr, Durham, North Carolina
  - East Carolina Univ School of Medicine, Greenville, North Carolina
  - Bowman Gray School of Medicine, Winston-Salem, North Carolina
  - Case Western Reserve Univ, Cleveland, Ohio
  - Pennsylvania State Univ / Hershey Med Ctr, Hershey, Pennsylvania
  - Univ TX Galveston Med Branch, Galveston, Texas